CLINICAL TRIAL: NCT02908867
Title: Therapeutic Strategies in Sexual Function of Men With Spinal Cord Injury
Brief Title: Therapeutic Strategies in Sexual Function
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Josepha Karinne de Oliveira Ferro, Master degree, Universidade Federal de Pernambuco
Other Study IDs: THERAPEUTIC STRATEGIES SCI
Record Dates: First submitted 2016-09-18; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Male Sexual Dysfunction; Spinal Cord Injury
Keywords: Sexuality; Spinal cord injuries; Complementary Therapies; Medicinal plants
MeSH Terms: conditions — Spinal Cord Injuries; Sexuality

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Therapeutic strategies group: To know the main therapeutic strategies used by men with spinal cord injury in sexual dysfunctions, mainly medicinal plants.
  Interventions: Other: Therapeutic Strategies

INTERVENTIONS:
Other: Therapeutic Strategies — Using questionnaires (Erectile Function of International Index and American Impairment Scale) and search in public markets using semi structured form

SUMMARY:
Objectives: To know the main therapeutic strategies used by men with spinal cord injury in sexual dysfunctions.

DETAILED DESCRIPTION:
Methods: This is a descriptive observational study involving 24 men with a mean age of 32.62 (CI 28.65 to 36.60), with spinal cord injury, recruited in reference services in spinal cord injury Recife (PE). The subjects underwent neurological evaluation in accordance with the guidelines of the International Standards for Neurological Examination and Functional classification of Spinal Cord Injury (ISNCSCI), the American Spinal Injury Association (ASIA), assessment of sexual function through the Erectile Function of International Index (IIEF) and answered a semi-structured form to identify therapeutic strategies used in sexual function. To collect information about medicinal plants, a search was made in the surroundings of public markets located in the Metropolitan Region of Recife (PE).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of traumatic spinal cord injury
* injury time less than six months
* heterosexual
* sexually active

Exclusion Criteria:

* patients who had erectile dysfunction attributed to endocrine or metabolic disease order
* those who underwent surgery in the genital area, such as radical prostatectomy or penile implant
* cognitive impairment

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study involving 24 men with spinal cord injury, recruited in reference services in spinal cord injury Recife (PE). Aged between 18 and 60 years with a clinical diagnosis of traumatic spinal cord injury, injury time less than six months, heterosexual and sexually active. The study excluded patients who had erectile dysfunction attributed to endocrine or metabolic disease order, those who underwent surgery in the genital area, such as radical prostatectomy or penile implant and cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Therapeutic Strategies | one day
  Therapeutic Strategies assessed by semi structured form in public market

SECONDARY OUTCOMES:
level of neurological lesion | one day
  Level of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Degree of lesion | one day
  Degree of neurological lesion assessed by ASIA Impairment Scale (AIS) according to the International Standards for Neurological and Functional Examination Classification of Spinal Cord Injury
Male sexual dysfunction | one day
  Male Sexual Dysfunction assessed by International Index of Erectile Function (IIEF)

CONTACTS AND LOCATIONS:
Overall Officials: Josepha KO Ferro, master, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Josepha Karinne de Oliveira Ferro, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No